CLINICAL TRIAL: NCT01484288
Title: Baroreflex Activation Therapy in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 360025
Record Dates: First submitted 2011-11-29; First posted 2011-12-02 (Estimated); Results first posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Device group (Experimental): Barostim Neo system
  Interventions: Device: Barostim Neo System

INTERVENTIONS:
Device: Barostim Neo System — Baroreflex Activation Therapy using the Barostim Neo System
  Other Names: XR-1 System; Neo system

SUMMARY:
The purpose of this clinical investigation is to evaluate the efficacy and safety of the CVRx Barostim Neo System in the treatment of patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 21 years
* Symptomatic heart failure despite optimal, stable pharmacological therapy for at least 4 weeks

Exclusion Criteria:

* Significant carotid plaque or stenosis
* Known or suspected baroreflex failure or autonomic neuropathy
* Myocardial infarction, unstable angina, syncope, cerebral vascular accident, SCD, or received defibrillation therapy within the past 3 months
* Heart failure secondary to a reversible condition

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo G Gronda, MD, FESC, Principal Investigator — MultiMedica
Locations (1):
- MultiMedica, Milan, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 12 subjects enrolled, 1 subject was a screen failure and was not implanted.
Period: Overall Study
Arm/Group | Device Group
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Device Group
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
  Black/African Descent | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 11
York Heart Association (NYHA) Class III [Count of Participants; unit: Participants] — NYHA classification places patients in one of four categories based on how much they are limited during physical activity, where Class I indicates no limitation of physical activity and Class IV indicates the patient is unable to carry on any physical activity without discomfort. The patient has symptoms of heart failure at rest, and if any physical activity is undertaken, discomfort increases.
  Participants | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26 (5)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 118 (14)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 70 (9)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 72 (8)
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: Percentage of LVEF] | 31 (7)
B-type natriuretic peptide (BNP) [Mean (Standard Deviation); unit: pg/mL] | 314 (307)
6-Minute Hall Walk [Mean (Standard Deviation); unit: Meters] — The 6-Minute Hall Walk test is a measure of physical function by measuring the distance a patient can walk in a 6-minute time period.
  Meters | 304 (50)
Quality of Life (Minnesota Living with Heart Failure) [Mean (Standard Deviation); unit: units on a scale] — The Minnesota Living with Heart Failure Questionnaire is a 21-item questionnaire designed as a measure of heart failure, as indicated by its adverse effects on patients' lives. Each item is scored in a 6-point Likert Scale (0 to 5); therefore, the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life.
  units on a scale | 33 (30)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Sympathetic Nervous System Activity (MSNA Bursts/Min)
Description: Change in muscle sympathetic nerve activity (MSNA) in bursts/min at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Error); unit: bursts/min
Arm/Group | Device Group
Number analyzed (Participants) | 11
bursts/min | -13.8 (1.4)

2. Primary Outcome: Changes in Sympathetic Nervous System Activity (MSNA Bursts/100 Heartbeats)
Description: Changes in Muscle Sympathetic Nerve Activity (bursts/100 heartbeats) at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Error); unit: bursts/100 heartbeats
Arm/Group | Device Group
Number analyzed (Participants) | 11
bursts/100 heartbeats | -22.5 (2.5)

3. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Device Group
Number analyzed (Participants) | 11
mmHg | 0.2 (4.6)

4. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Device Group
Number analyzed (Participants) | 11
mmHg | -2.3 (2.6)

5. Secondary Outcome: Change in Heart Rate
Description: Change in heart rate at 6 months compared to baseline
Time Frame: 6 months
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Device Group
Number analyzed (Participants) | 11
bpm | -0.2 (3.0)

6. Secondary Outcome: Change in Six-Minute Hall Walk
Description: Change in six-minute hall walk distance at 6 months compared to baseline. The 6-Minute Hall Walk test is a measure of physical function by measuring the distance a patient can walk in a 6-minute time period.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Meters
Arm/Group | Device Group
Number analyzed (Participants) | 11
Meters | 51.1 (25.6)

7. Secondary Outcome: New York Heart Association (NYHA) Class
Description: Number of patients with NYHA Class I-IV at 6 months. NYHA classification places patients in one of four categories based on how much they are limited during physical activity, where Class I indicates no limitation of physical activity and Class IV indicates the patient is unable to carry on any physical activity without discomfort. The patient has symptoms of heart failure at rest, and if any physical activity is undertaken, discomfort increases.
Time Frame: Six months
Population: NYHA Class was not available for 1 patient at the 6-month timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Device Group
Number analyzed (Participants) | 10
Participants
  Class I | 9
  Class II | 1
  Class III | 0
  Class IV | 0

8. Secondary Outcome: Change in Quality of Life (Minnesota Living With Heart Failure Questionnaire)
Description: Change in Quality of Life as measured by the Minnesota Living with Heart Failure Questionnaire at 6 months compared to baseline.
  The Minnesota Living with Heart Failure Questionnaire is a 21-item questionnaire designed as a measure of heart failure, as indicated by its adverse effects on patients' lives. Each item is scored in a 6-point Likert Scale (0 to 5); therefore, the total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of life.
Time Frame: Six months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Device Group
Number analyzed (Participants) | 11
units on a scale | -10.6 (3.8)

9. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF)
Description: Change in LVEF at 6 months compared to baseline
Time Frame: Six months
Measure: Mean (Standard Error); unit: percentage of LVEF
Arm/Group | Device Group
Number analyzed (Participants) | 11
percentage of LVEF | 0.8 (1.9)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Device Group
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 7/11
Other Adverse Events (participants affected / at risk) | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Group (N=11)
Acute decompensated heart failure (Cardiac disorders) | 3 (4)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Gallstones (Hepatobiliary disorders) | 1 (1)
Epididymo-orchitis (Infections and infestations) | 1 (1)
Tremor aggravated (Nervous system disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device Group (N=11)
supraventricular tachycardia (Cardiac disorders) | 1 (1)
Diabetic foot ulcer (Endocrine disorders) | 1 (2)
Epistaxis (Vascular disorders) | 1 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No